CLINICAL TRIAL: NCT05491603
Title: An Observer-Blinded, Randomized, Aqueous Gel-Controlled Trial of the Safety and Efficacy of DBI-001 Gel, DBI-002 Gel, and Aqueous Gel in Subjects With Onychomycosis
Brief Title: A Trial to Evaluate the Safety and Efficacy of DBI-001 Gel, DBI-002 Gel, and Aqueous Gel in Subjects With Onychomycosis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Suspended: Study halted prematurely but potentially will resume. Sponsor suspension, and not due to safety or site-related matters.
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-206
Record Dates: First submitted 2022-07-28; First posted 2022-08-08 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-02

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — BANG polymer gel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DBI-001 Gel (Experimental): Topical application of DBI-001 gel on foot/feet affected with onychomycosis.
  Interventions: Biological: DBI-001
- DBI-002 Gel (Experimental): Topical application of DBI-002 gel on foot/feet affected with onychomycosis.
  Interventions: Biological: DBI-002
- Aqueous Gel (Placebo Comparator): Topical application of aqueous gel on foot/feet affected with onychomycosis.
  Interventions: Biological: Aqueous Gel

INTERVENTIONS:
Biological: DBI-001 — Topically administered
  Arms: DBI-001 Gel
Biological: DBI-002 — Topically administered
  Arms: DBI-002 Gel
Biological: Aqueous Gel — Topically administered
  Arms: Aqueous Gel

SUMMARY:
This is a randomized, observer-blinded, Aqueous Gel-controlled trial examining the safety and efficacy of daily application of DBI-001 Gel vs. DBI-002 Gel vs. Aqueous Gel for 24 consecutive weeks in subjects with onychomycosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age, inclusive, at Screening
* Willing to abstain from all cosmetic activities involving the toenails during the entire course of the study
* Distal subungual onychomycosis defined as a great toenail with onycholysis and thickening of the nail bed with keratinous material
* Willing to have his/her treatment-targeted great toenail(s) clipped to remove onycholytic nail plate at each visit
* At least one treatment-targeted great toenail must have at least 6 mm of clear nail from the proximal nail fold to the proximal limit of disease and, after trimming to within 1mm distal nail groove, have at least 3mm of involved nail from distal nail groove to proximal limit of disease
* Confirmed presence of microorganisms of interest by KOH and qPCR at Screening
* The affected treatment-targeted great toenail(s) is capable of re-growth as documented by subject self-reported history of clipping nails at least monthly

Exclusion Criteria:

* Positive urine pregnancy test, pregnant, lactating, or female of childbearing potential who does not agree to use an active method of birth control for the duration of the study
* Any dermatological conditions that could interfere with clinical evaluations
* Great toenails with only superficial white onychomycosis, any evidence of subungual mycetoma as evidenced by yellow or white spikes, or any evidence of proximal onychomycosis
* Any underlying disease(s) or other dermatological condition(s) that requires the use of interfering topical or systemic therapy, with the exception of certain protocol-specified that require a defined washout period for eligibility
* Treatment of any type of cancer within the last 6 months, with the exception of superficial skin cancers such as basal cell carcinoma and squamous cell carcinoma
* History of any significant internal disease which contraindicates the use of live microbiome
* History of failing oral or prescription topical treatment for onychomycosis
* A history of current episode of onychomycosis present for more than 3 years
* Nail or anatomic abnormalities of the target great toenail(s)
* AIDS or AIDS-related complex by medical history
* History of current street drug or alcohol abuse, or street drug or alcohol abuse within the past year
* Subjects known or suspected to be taking immune suppressive medications or subjects who are immunosuppressed
* Subjects with poorly controlled diabetes mellitus requiring medical intervention/treatment
* Subjects with peripheral vascular disease based on medical history
* Subjects who have participated in any other trial of an investigational drug or device within 60 days prior to enrollment or participation in a research study concurrent with this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of involved great toenail(s) | 24 weeks of participation
  Absolute change from Baseline in percent of involved treatment-targeted great toenail(s) at Week 24.
Changes in signs and symptoms of Onychomycosis | Baseline through End of Study (up to 48 weeks of participation)
  Change from baseline in individual signs and symptoms at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48 of sites treated with DBI-001 Gel or DBI-002 Gel. The minimum value is 0 and the maximum value is 4.

SECONDARY OUTCOMES:
Change in percentage of involved great toenail(s) | 48 weeks of participation
  Absolute change from Baseline in percent of involved treatment-targeted great toenail(s) at Week 48.
Population with completely clear nail growth | 48 weeks of participation
  Proportion of subjects with completely clear nail growth of the treatment-targeted great toenail(s) at Weeks 24 and 48 based on measurements from digital images.
Change in Investigator's Static Global Assessment (ISGA) | 48 weeks of participation
  Change from Baseline in Investigator's Static Global Assessment (ISGA) for the treatment-targeted great toenail(s) at Weeks 24 and 48. The minimum value of ISGA is 0 and the maximum value is 4.
Length of new clear nail growth | 48 weeks of participation
  Length in mm of new clear nail growth based on measurements from digital images at Weeks 24 and 48 of treatment-targeted great toenail(s).
Molecular diagnostic quantitative polymerase chain reaction (qPCR) and whole genome sequencing (WGS) comparison of DBI-001 Gel, DBI-002 Gel and Aqueous Gel on the impact of T. rubrum levels | 48 weeks of participation
  Antimicrobial efficacy and microbiome community analysis
Change in colony forming units after using DBI-001 Gel or DBI-002 Gel or Aqueous Gel at Weeks 24 and 48 | 48 weeks of participation
  Antimicrobial efficacy
Evaluate the presence of DBI-001, DBI-002 based on qPCR and WGS and Weeks 24 and 48 | 48 weeks of participation
  Antimicrobial efficacy and microbiome community analysis
Evaluate the effect of DBI-001 Gel and DBI-002 Gel on the change in relative abundance and diversity of the cutaneous microbiome of the great toenail(s) from Screening to Weeks 24 and 48 as measured by WGS | 48 weeks of participation
  Antimicrobial efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Emma Taylor, M.D., Study Director — DermBiont, Inc.
Locations (5):
- United States (5):
  - T. Joseph Raoof MD, Inc./Encino Research Center, Encino, California
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Oregon Dermatology and Research Center, Portland, Oregon
  - DermResearch, Austin, Texas
  - North Sound Dermatology, Mill Creek, Washington